CLINICAL TRIAL: NCT04941794
Title: Biomarkers as Predictors of Chronic Heart Failure in Patients With Type 2 Diabetes
Status: Recruiting | Type: Observational
Sponsor: Regionshospital Nordjylland (Other Government)
Responsible Party: Sponsor
Other Study IDs: N-20210021
Record Dates: First submitted 2021-06-21; First posted 2021-06-28 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Type 2 Diabetes; Chronic Heart Failure
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A cohort study on patients with type 2 diabetes to investigate possible biomarkers as predictors of chronic heart failure.

DETAILED DESCRIPTION:
A cohort study on 500 patients with type 2 diabetes without known heart disease and age > 50 years of age. On inclusion and on yearly basis, patients are evaluated by echocardiography, ECG, blood tests to examine NT-ProBNP, hs-CRP, troponin, kidney function and 6 minutes hall walk test.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* age > 50 years

Exclusion Criteria:

* History of acute or chronic heart failure
* History of ischemic heart disease

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 500 patients with known type 2 diabetes who are treated at the department of endocrinology, North Denmark Regional Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Chronic Heart Failure | During 5 year follow up
  Determined by echocardiography according to European Society of Cardiology (ESC) definitions

SECONDARY OUTCOMES:
NT-ProBNP | During 5 year follow up
  Change in N-terminal prohormone of brain natriuretic peptide (NT-ProBNP)
hs-CRP | During 5 year follow up
  Change in High-sensitivity C-reactive protein (hs-CRP)
Troponin | During 5 year follow up
  Change in Troponin
6 minutes walk test | During 5 year follow up
  Change in 6 minutes walk test

OTHER OUTCOMES:
HOMA-IR | During 5 year follow-up
  Change in Homeostatic Model Assessment for Insulin Resistance (HOMA-IR)

CONTACTS AND LOCATIONS:
Overall Officials: Steen Hylgaard Jørgensen, MD, Principal Investigator — Department of Cardiology
Locations (1):
- North Denmark Regional Hospital, Hjørring, Denmark